CLINICAL TRIAL: NCT02965781
Title: A Phase 2, Multi-site, Randomized, Double-blind, Vehicle-controlled Study of the Efficacy and Safety of Squaric Acid Dibutyl Ester (SADBE) in Subjects With Recurrent Herpes Labialis - Single Versus Two-dose Arm Application
Brief Title: Double-blind, Vehicle-controlled Study of the Efficacy and Safety of SADBE in Subjects With Recurrent Herpes Labialis
Acronym: P2a
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Squarex, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P2a
Record Dates: First submitted 2016-10-24; First posted 2016-11-17 (Estimated); Results first posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Herpes Labialis; Cold Sore
MeSH Terms: conditions — Herpes Labialis | interventions — squaric acid dibutyl ester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- One SADBE application (Active Comparator): Patient will receive a topical 2% SADBE sensitization dose applied to the patient's upper arm. Three weeks after topical sensitization dose patient will receive topical placebo applied to the patient's upper arm.
  Interventions: Drug: SADBE; Other: Placebo
- Two SADBE applications (Active Comparator): Patient will receive a topical 2% SADBE sensitization dose applied to the patient's upper arm. A 0.5% SADBE intensification dose will be applied to the patient's upper arm 3 weeks after sensitization dose.
  Interventions: Drug: SADBE
- Placebo application (DMSO only-No SADBE) (Placebo Comparator): Patient will receive a topical placebo (vehicle-DMSO) dose applied to the patient's upper arm. A topical placebo (vehicle-DMSO) follow up dose will be applied to the patient's upper arm 3 weeks after the first placebo dose dose.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SADBE — Topical solution
  Other Names: Squaric acid dibutyl ester
  Arms: One SADBE application; Two SADBE applications
Other: Placebo — Topical solution
  Other Names: Vehicle-DMSO
  Arms: One SADBE application; Placebo application (DMSO only-No SADBE)

SUMMARY:
This study evaluates the safety and efficacy of SADBE in the prevention of recurrent herpes labialis in adults. Two-thirds of the participants will receive a SADBE solution, while the other third will receive only the vehicle as a placebo control. The solutions will be administered topically to the patient's arms. The study will compare a single-arm application versus a two-arm application versus two placebo doses on the arm.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Clinical diagnosis of herpes labialis, which may be made at the screening visit based on the patient's self-reported history of symptoms. An active herpes labialis outbreak at the time of entry into the clinical trial will neither be required nor will be an exclusion criteria.
* Self report having four or more episodes of herpes labialis in the past 12 months

Exclusion Criteria:

* People that have had treatment with anti viral therapy within 2 weeks before sensitization dose.
* Pregnant or lactating females.
* Current or recurrent non-herpetic infection or any underlying condition that may predispose to infection or anyone who has been admitted to the hospital due to bacteremia, pneumonia or any other serious infection.
* Therapy with glucocorticoid or immunosuppressants at time of recruitment or within past 4 weeks, except for inhaled corticosteroids for asthma or topical steroids in sites other than face.
* History of malignancy (except patients with surgically cured basal cell or squamous cell skin cancers)
* History of organ transplantation
* HIV-positive status determined by history at screening or known history of any other immunosuppressive disease.
* Severe co-morbidities (diabetes mellitus requiring insulin, CHF (EF<50% at baseline will be exclusionary) MI, CVA or TIA within 3 months of screening visit, unstable angina pectoris, oxygen-dependent severe pulmonary disease
* History of exposure to squaric acid or squaric acid dibutyl ester.
* Known hypersensitivity to DMSO
* Any condition judged by the investigator to cause this clinical trial to be detrimental to the patient.
* Subject is currently enrolled in another investigational device or drug trial(s), or subject has received other investigational agent(s) within 28 days of baseline visit.
* Previous or current participation in a clinical trial of SADBE to treat herpes labialis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugh McTavish, PhD, JD, Study Director — Squarex, LLC; Thomas D Horn, MD, Study Chair — Squarex, LLC
Locations (5):
- United States (5):
  - Stanford Medicine Outpatient Center, Redwood City, California
  - International Research Partners, LLC, Doral, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Quality Clinical Research, Inc, Omaha, Nebraska
  - Advantage Clinical Trials, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | One SADBE Application | Two SADBE Applications | Placebo Application (DMSO Only-No SADBE)
Started | 46 | 46 | 47
Completed | 46 | 46 | 47
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | One SADBE Application | Two SADBE Applications | Placebo Application (DMSO Only-No SADBE) | Total
Number analyzed (Participants) | 46 | 46 | 47 | 139
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 46 | 46 | 47 | 139
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 47.8 [19.8 to 82.6] | 44.2 [23.8 to 80.4] | 50.1 [21.1 to 82.6] | 47.1 [19.8 to 82.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 28 | 26 | 85
  Male | 15 | 18 | 21 | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 2 | 1 | 4
  Black | 11 | 7 | 8 | 26
  Hispanic | 13 | 18 | 17 | 48
  White | 21 | 18 | 21 | 60
  Unasnswered | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 46 | 46 | 47 | 139
HSV-1-neg / HSV-2 neg [Count of Participants; unit: Participants] | 1 | 2 | 3 | 6
HSV-1-neg / HSV-2 pos [Count of Participants; unit: Participants] | 1 | 3 | 5 | 9
HSV-1-pos / HSV-2 neg [Count of Participants; unit: Participants] | 30 | 19 | 24 | 73
HSV-1-pos / HSV-2 pos [Count of Participants; unit: Participants] | 14 | 22 | 13 | 49
Median self-reported prior outbreaks over 12 months [Count of Participants; unit: Participants] | 6 | 6 | 6 | 18
4 or 5 prior outbreaks [Count of Participants; unit: Participants] | 19 | 15 | 21 | 55
6 or more prior outbreaks [Count of Participants; unit: Participants] | 27 | 31 | 25 | 83

OUTCOME MEASURES:

1. Primary Outcome: Days to Next Herpes Labialis (Cold Sore) Episode From 43 Days After the First Dose up to 121 Days After the First Dose
Description: The number of days until a patient reports his or her first new herpes labialis episode from 43 - 121 days following the first dose
Time Frame: 43 - 121 days after the first dose
Measure: Median (Full Range); unit: days
Groups:
- Placebo Application (DMSO Only-No SADBE): Placebo
- Two SADBE Applications: 2-dose
- One SADBE Application: 1-dose
Arm/Group | Placebo Application (DMSO Only-No SADBE) | Two SADBE Applications | One SADBE Application
Number analyzed (Participants) | 43 | 44 | 41
days | 128 [4 to 318] | 163 [7 to 318] | 174 [17 to 318]

2. Secondary Outcome: Number of Outbreaks Beginning 43 Days After the First Dose up to 12 Months
Description: The number of new herpes labialis episodes per subject during the 12-month follow up period following the first drug dose, beginning day 43 after the first dose
Time Frame: From day 43 after the first dose up to 12 months
Measure: Mean (Standard Deviation); unit: outbreaks per participant
Arm/Group | Placebo Application (DMSO Only-No SADBE) | Two SADBE Applications | One SADBE Application
Number analyzed (Participants) | 43 | 44 | 41
outbreaks per participant | 0.610 (0.802) | 0.500 (0.849) | 0.231 (0.427)

ADVERSE EVENTS:
Time Frame: 1 Year
Description: Subjects receiving One or Two doses of SADBE were combined for Adverse Event Reporting because they did not experience adverse events at different incidence rates.
  The terms mild, moderate, and severe were undefined except "severe" was defined as requiring topical corticosteroid treatment and none of these events correspond to a serious adverse event or to Common Terminology Criteria for Adverse Events (CTCAE) v 5.0 terms for skin and subcutaneous tissue disorders.
Arm/Group | Placebo Application (DMSO Only-No SADBE) | Two SADBE Applications | One SADBE Application
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/46 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 17/47 | 19/46 | 18/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Application (DMSO Only-No SADBE) (N=47) | Two SADBE Applications (N=46) | One SADBE Application (N=46)
Dead skin at application site (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis at application site (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Erythema, stain, or rash at application site (Skin and subcutaneous tissue disorders) | 4 | 7 | 6
Erythema distal from application site (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Flushed burning sensation on face (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Herpes lesion on genitals, anus, or spine (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Irritation, itching at application site (Skin and subcutaneous tissue disorders) | 1 | 3 | 4
Irritation, itching distal from application site (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Lightheadedness (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pimple (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Purpura at application site (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Papule on lip (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis from adhesive (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Burning at application site. (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Tingling, stinging at application site (Skin and subcutaneous tissue disorders) | 4 | 0 | 0
Tingling distal from application site (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Boil at application site (Skin and subcutaneous tissue disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-16): https://cdn.clinicaltrials.gov/large-docs/81/NCT02965781/Prot_SAP_000.pdf